CLINICAL TRIAL: NCT00316407
Title: Phase I/II Lapatinib Plus Carboplatin and Paclitaxel in Stage III or IV Relapsed Ovarian or Stage IV Breast Cancer Patients
Brief Title: Lapatinib/Carboplatin/Paclitaxel in Previously Treated Ovarian or Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Saul Rivkin, M.D., Swedish Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC 0503
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2010-03

CONDITIONS: Ovarian Epithelial Cancer Stage III; Stage IV Ovarian Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms; Breast Neoplasms | interventions — Lapatinib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lapatinib (GW572016) — 1000 mg po qd
  Other Names: Tykerb
Drug: Carboplatin — AUC 2 weekly x 3 of 4 week cycle
  Other Names: Paraplatin
Drug: Paclitaxel — 60 mg/m2 weekly x 3 of 4 week cycle
  Other Names: Taxol

SUMMARY:
The purpose of this study is to determine the effectiveness, safety, tolerability and best dose of Lapatinib (GW572016) in combination with carboplatin and paclitaxel.

DETAILED DESCRIPTION:
The MTD was found in the phase I portion of this study to be oral lapatinib 1000 mg per day for each 4 week cycle and paclitaxel 60 mg/m2 weekly x 3 of a 4 week cycle and carboplatin AUC 2 weekly x 3 of a 4 week cycle.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed (Stage III or IV) ovarian, primary peritoneal, fallopian tube carcinoma patients.
* Stage IV metastatic breast cancer patients who have failed no more than four previous chemotherapies for Stage IV disease.
* Ability to swallow and retain oral medications.
* Measurable disease

Exclusion Criteria:

* Treatment with previous weekly carboplatin and paclitaxel.
* No prior treatment with erbB targeting therapies such as erlotinib, gefitinib and cetuximab.
* No concomitant requirement for medication classification as CYP3A4 inducers or inhibitors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Toxicity | 1 year

SECONDARY OUTCOMES:
Objective response (PR or CR) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Saul Rivkin, MD, Principal Investigator — Swedish Medical Center Cancer Institute
Locations (2):
- United States (2):
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Swedish Medical Center Cancer Institute, Seattle, Washington